CLINICAL TRIAL: NCT00789477
Title: A Double-Masked, Randomized, Controlled Study of the Safety, Tolerability and Biological Effect of Repeated Intravitreal Administration of VEGF Trap-Eye in Patients With Diabetic Macular Edema (DME)
Brief Title: DME And VEGF Trap-Eye [Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321)] INvestigation of Clinical Impact
Acronym: DA VINCI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VGFT-OD-0706
Record Dates: First submitted 2008-11-07; First posted 2008-11-11 (Estimated); Results first posted 2014-09-09 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-08

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Intravitreal Aflibercept Injection .5Q4 (Experimental): Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) .5 mg every 4 weeks
  Interventions: Drug: Intravitreal Aflibercept Injection
- Intravitreal Aflibercept Injection 2Q4 (Experimental): Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2 mg every 4 weeks
  Interventions: Drug: Intravitreal Aflibercept Injection
- Intravitreal Aflibercept Injection 2Q8 (Experimental): Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2mg every 4 weeks for 3 visits followed by every 8 weeks
  Interventions: Drug: Intravitreal Aflibercept Injection
- Intravitreal Aflibercept Injection 2PRN (Experimental): Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2mg every 4 weeks for 3 visits followed by PRN (as-needed) dosing according to the re-treatment criteria
  Interventions: Drug: Intravitreal Aflibercept Injection
- Laser Photocoagulation (Active Comparator): Focal laser at week 1, and one week after visits at which the participant met laser re-treatment criteria to the end of the study (week 52) starting at week 16; laser re- treatment was permitted no more than once every 16 weeks.
  Interventions: Procedure: Laser Photocoagulation

INTERVENTIONS:
Procedure: Laser Photocoagulation — laser every 16 weeks as needed
  Other Names: macular laser therapy
  Arms: Laser Photocoagulation
Drug: Intravitreal Aflibercept Injection
  Other Names: IAI; EYLEA®; BAY86-5321; VEGF Trap-Eye
  Arms: Intravitreal Aflibercept Injection .5Q4; Intravitreal Aflibercept Injection 2PRN; Intravitreal Aflibercept Injection 2Q4; Intravitreal Aflibercept Injection 2Q8

SUMMARY:
This is a Phase 2, doubled-masked, randomized study of the efficacy and safety of Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) in subjects with diabetic macular edema (DME). Approximately 200 subjects will be randomized in the US, Canada, Australia and EU.

DETAILED DESCRIPTION:
Qualified subjects will be randomized to one of 5 treatment arms. The active (treatment) phase of the study will be 52 weeks, with a 6 month safety follow-up

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinically significant DME with central involvement
* Adults 18 years or older with type 1 or 2 diabetes mellitus with diabetic macular edema
* ETDRS BCVA: 20/40 to 20/320 (letter score of 73 to 24) in the study eye

Exclusion Criteria:

* History of vitreoretinal surgery in the study eye
* Panretinal laser photocoagulation or macular laser photocoagulation in the study eye within 3 months of screening
* Previous use of intraocular or periocular corticosteroids in the study eye within 3 months of screening
* Previous treatment with anti-angiogenic drugs in either eye (pegaptanib sodium, anecortave acetate, bevacizumab, ranibizumab, etc) within 3 months of screening
* Uncontrolled diabetes mellitus
* Uncontrolled hypertension defined as systolic > 180mmHg or > 160 mmHg on 2 consecutive measurements or diastolic > 100 mmHg on optimal medical regimen
* Ocular disorders in the study eye, other than DME, that may confound interpretation of study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2008-12; Primary Completion 2009-12 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (46):
- United States (41):
  - Artesia, California
  - Beverly Hills, California
  - Mountain View, California
  - Pasadena, California
  - Sacramento, California
  - Santa Ana, California
  - Hamden, Connecticut
  - New London, Connecticut
  - Boynton Beach, Florida
  - Fort Lauderdale, Florida
  - Fort Myers, Florida
  - Ocala, Florida
  - Palm Beach Gardens, Florida
  - Winter Haven, Florida
  - Augusta, Georgia
  - Honolulu, Hawaii
  - Indianapolis, Indiana
  - Bangor, Maine
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Jackson, Michigan
  - Kansas City, Missouri
  - Lincoln, Nebraska
  - New Brunswick, New Jersey
  - Northfield, New Jersey
  - Toms River, New Jersey
  - Rochester, New York
  - Charlotte, North Carolina
  - Raleigh, North Carolina
  - Cincinnati, Ohio
  - Pittsburgh, Pennsylvania
  - Greenville, South Carolina
  - West Columbia, South Carolina
  - Nashville, Tennessee
  - Abilene, Texas
  - Arlington, Texas
  - Austin, Texas
  - Houston, Texas
  - McAllen, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
- Vienna, Austria
- Canada (4):
  - Vancouver, British Columbia
  - Victoria, British Columbia
  - London, Ontario
  - Mississauga, Ontario

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 221 participants were randomized at 39 sites in the US, Canada, and Austria. After the 1 year treatment period, participants were to be followed for safety in a 6 mo. follow-up phase. The last visit for this study occurred in September, 2010.
Pre-assignment Details: The study population consisted of men and women aged 18 or older with clinically significant diabetic macular edema (DME) with central involvement, and a best corrected visual acuity (BCVA) of 20/40 to 20/320 (letter score of 73 to 24) in the study eye.
Groups:
- Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321).5Q4: Intravitreal Aflibercept Injection (IAI) 0.5 mg every 4 weeks to week 52
- Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2Q4: Intravitreal Aflibercept Injection (IAI) 2 mg every 4 weeks to week 52
- Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2Q8: Intravitreal Aflibercept Injection (IAI) 2mg every 4 weeks for 3 visits followed by every 8 weeks through week 52
- Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321)2PRN: Intravitreal Aflibercept Injection (IAI) 2mg every 4 weeks for 3 visits followed by PRN (as-needed) dosing according to the re-treatment criteria to week 52
Period: Overall Study
Arm/Group | Laser Photocoagulation | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321).5Q4 | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2Q4 | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2Q8 | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321)2PRN
Started | 44 (randomized) | 44 (randomized) | 44 (randomized) | 44 (randomized) | 45 (randomized)
Participants Received Treatment | 44 (safety analysis set (SAF)) | 44 (SAF) | 44 (SAF) | 42 (SAF) | 45 (SAF)
Completed | 33 | 38 | 33 | 34 | 38
Not Completed | 11 | 6 | 11 | 10 | 7
Not completed — Withdrawal by Subject | 2 | 1 | 3 | 2 | 3
Not completed — Protocol Violation | 1 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 3 | 3 | 1 | 0 | 0
Not completed — Death | 1 | 1 | 2 | 2 | 0
Not completed — Lost to Follow-up | 0 | 1 | 4 | 2 | 4
Not completed — Lack of Efficacy | 2 | 0 | 0 | 0 | 0
Not completed — Other | 2 | 0 | 1 | 3 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS): included all randomized patients who received any study drug, had baseline assessments, and had at least one (1) post-baseline assessment.
Groups:
- Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321).5Q4: Intravitreal Aflibercept Injection (IAI) 0.5mg every 4 weeks to week 52
- Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2Q4: Intravitreal Aflibercept Injection (IAI) 2mg every 4 weeks to week 52
- Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321)2PRN: Intravitreal Aflibercept Injection (IAI) 2mg every 4 weeks for 3 visits followed by PRN dosing according to the re-treatment criteria to week 52
- Total: Total of all reporting groups
Arm/Group | Laser Photocoagulation | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321).5Q4 | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2Q4 | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2Q8 | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321)2PRN | Total
Number analyzed (Participants) | 44 | 44 | 44 | 42 | 45 | 219
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.0 (8.12) | 62.3 (10.70) | 62.1 (10.50) | 62.5 (11.49) | 60.7 (8.66) | 62.3 (9.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 20 | 17 | 20 | 16 | 90
  Male | 27 | 24 | 27 | 22 | 29 | 129

OUTCOME MEASURES:

1. Primary Outcome: Change in BCVA From Baseline to Week 24 - Last Observation Carried Forward (LOCF)
Description: Visual function of the study eye was assessed using the Early Treatment Diabetic Retinopathy Study (ETDRS) protocol at 4 meters. Measurements were taken at every study visit.
  Missing values were imputed with post-baseline values during on-treatment period by using last observation carried forward (LOCF).
Time Frame: At week 24
Population: The FAS was used for the primary efficacy analysis. It included patients as randomized.
Measure: Mean (Standard Deviation); unit: letters correctly read
Groups:
- Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2Q4: Intravitreal Aflibercept Injection (IAI) 2mg every 4 weeks for 3 visits followed by every 8 weeks through week 52
- Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2Q8: Intravitreal Aflibercept Injection (IAI) 2mg every 4 weeks for 3 visits followed by every 8 weeks to week 52
Arm/Group | Laser Photocoagulation | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321).5Q4 | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2Q4 | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2Q8 | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321)2PRN
Number analyzed (Participants) | 44 | 44 | 44 | 42 | 45
letters correctly read | 2.5 (16.14) | 8.6 (14.64) | 11.4 (8.67) | 8.5 (7.50) | 10.3 (7.52)

2. Secondary Outcome: Change in BCVA From Baseline to Week 52 - LOCF
Description: Visual function of the study eye was assessed using the Early Treatment Diabetic Retinopathy Study (ETDRS) protocol at 4 meters. Missing values were imputed with post-baseline values during on-treatment period by using last observation carried forward (LOCF).
Time Frame: At week 52
Population: FAS
Measure: Mean (Standard Deviation); unit: letters correctly read
Arm/Group | Laser Photocoagulation | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321).5Q4 | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2Q4 | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2Q8 | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321)2PRN
Number analyzed (Participants) | 44 | 44 | 44 | 42 | 45
letters correctly read | -1.3 (20.72) | 11.0 (15.40) | 13.1 (10.54) | 9.7 (8.93) | 12.0 (11.09)

3. Secondary Outcome: Participants With Gains in ETDRS Letter Score of at Least 15 Letters - LOCF
Description: Missing values were imputed with post-baseline values during on-treatment period by using last observation carried forward (LOCF).
Time Frame: At week 24 and week 52
Population: FAS
Measure: Number; unit: participants
Arm/Group | Laser Photocoagulation | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321).5Q4 | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2Q4 | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2Q8 | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321)2PRN
Number analyzed (Participants) | 44 | 44 | 44 | 42 | 45
participants
  At week 24 | 9 (135.17) | 15 (110.65) | 14 (143.04) | 7 (141.78) | 12 (132.17)
  At week 52 | 5 | 18 | 20 | 10 | 19

4. Secondary Outcome: Change From Baseline in Central Retinal Thickness (CRT) as Assessed by Optical Coherence Tomography (OCT) - LOCF
Description: Retinal thickness was evaluated using OCT at every visit except week 1. Missing values were imputed with post-baseline values during on-treatment period by using last observation carried forward (LOCF).
Time Frame: At week 24 and week 52
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | Laser Photocoagulation | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321).5Q4 | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2Q4 | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2Q8 | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321)2PRN
Number analyzed (Participants) | 43 | 44 | 44 | 42 | 45
microns
  At week 24 | -67.9 (135.17) | -144.6 (110.65) | -194.5 (143.04) | -127.3 (141.78) | -153.3 (132.17)
  At week 52 | -58.4 (177.60) | -165.4 (135.72) | -227.4 (148.96) | -187.8 (135.01) | -180.3 (124.43)

5. Secondary Outcome: Number of Focal Laser Treatments
Time Frame: Week 1 to week 48
Population: For the first 24 weeks, the Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) groups did not receive laser treatment. From week 24 onward, participants in the Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) groups were allowed to receive laser rescue treatment.
Measure: Mean (Standard Deviation); unit: Treatments
Arm/Group | Laser Photocoagulation | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321).5Q4 | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2Q4 | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2Q8 | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321)2PRN
Number analyzed (Participants) | 44 | 44 | 44 | 42 | 45
Treatments | 2.5 (0.87) | 0.8 (0.93) | 0.5 (0.66) | 0.8 (0.86) | 0.7 (0.77)

ADVERSE EVENTS:
Time Frame: Day 1 to week 52
Description: Safety analysis set (SAF): included all patients who received any study drug. The SAF was used for all safety and tolerability assessments. Safety analysis included patients as treated.
Arm/Group | Laser Photocoagulation | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321).5Q4 | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2Q4 | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2Q8 | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321)2PRN
Serious Adverse Events (participants affected / at risk) | 10/44 | 14/44 | 13/44 | 12/42 | 6/45
Other Adverse Events (participants affected / at risk) | 20/44 | 22/44 | 22/44 | 26/42 | 24/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Laser Photocoagulation (N=44) | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321).5Q4 (N=44) | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2Q4 (N=44) | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2Q8 (N=42) | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321)2PRN (N=45)
Abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 2 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Angle closure glaucoma (Eye disorders) | 0 | 0 | 1 | 0 | 0 — Study eye
Aortic stenosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Blood pressure increased (Investigations) | 0 | 1 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Cardiac failure acute (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 3 | 1 | 2
Cellulitis (Infections and infestations) | 0 | 3 | 2 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 1 | 2 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 2 | 0 | 3
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Colon cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Corneal abrasion (Eye disorders) | 0 | 0 | 0 | 1 | 0 — Study eye
Coronary artery disease (Cardiac disorders) | 0 | 1 | 1 | 0 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 1 | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Cystoid macular oedema (Eye disorders) | 0 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0
Device occlusion (General disorders) | 0 | 1 | 0 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0
Diabetic retinal oedema (Eye disorders) | 1 | 0 | 0 | 0 | 0 — Study eye
Diabetic retinopathy (Eye disorders) | 0 | 0 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Endophthalmitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 — Study eye
Fluid overload (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0
Gangrene (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Hemiparesis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 2 | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Hypertensive emergency (Vascular disorders) | 1 | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Joint capsule rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 1 | 0 | 0
Localised infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Maculopathy (Eye disorders) | 0 | 0 | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0
Multi-organ failure (General disorders) | 0 | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 2 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Nephropathy (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Parotitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 1 | 0
Renal cell carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Retinal tear (Eye disorders) | 0 | 0 | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Sick sinus syndrome (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Silent myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Stress urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Sudden death (General disorders) | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Traumatic brain injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Uveitis (Eye disorders) | 0 | 1 | 0 | 0 | 0 — Study eye
Varices oesophageal (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Visual acuity reduced (Eye disorders) | 1 | 0 | 0 | 0 | 0
Visual acuity reduced (Eye disorders) | 1 | 0 | 0 | 0 | 0 — Study eye
Vitreous adhesions (Eye disorders) | 0 | 0 | 0 | 0 | 1
Vitreous haemorrhage (Eye disorders) | 3 | 0 | 0 | 0 | 0 — Study eye
Vitreous haemorrhage (Eye disorders) | 1 | 1 | 1 | 2 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Wolff-Parkinson-White syndrome (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Laser Photocoagulation (N=44) | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321).5Q4 (N=44) | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2Q4 (N=44) | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2Q8 (N=42) | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321)2PRN (N=45)
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 3 | 4 | 5
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 1
Blepharitis (Eye disorders) | 0 | 0 | 4 | 0 | 1
Blepharitis (Eye disorders) | 0 | 0 | 4 | 0 | 1 — Study eye
Blood glucose increased (Investigations) | 1 | 4 | 3 | 6 | 6
Blood potassium increased (Investigations) | 0 | 1 | 0 | 3 | 3
Blood pressure increased (Investigations) | 1 | 1 | 4 | 1 | 1
Blood urine present (Investigations) | 0 | 1 | 0 | 1 | 3
Bronchitis (Infections and infestations) | 1 | 3 | 2 | 0 | 2
Cataract (Eye disorders) | 1 | 2 | 1 | 0 | 5
Cataract (Eye disorders) | 2 | 2 | 3 | 2 | 5 — Study eye
Conjunctival haemorrhage (Eye disorders) | 8 | 12 | 7 | 15 | 13
Corneal abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 2 | 3 — Study eye
Diabetic retinal oedema (Eye disorders) | 0 | 4 | 3 | 0 | 4
Diabetic retinal oedema (Eye disorders) | 0 | 1 | 3 | 1 | 3 — Study eye
Eye pain (Eye disorders) | 3 | 2 | 0 | 1 | 0
Eye pain (Eye disorders) | 2 | 6 | 5 | 6 | 7 — Study eye
Foreign body sensation in eye (Eye disorders) | 0 | 1 | 1 | 1 | 3 — Study eye
Glucose urine present (Investigations) | 1 | 1 | 0 | 3 | 4
Glycosylated haemoglobin increased (Investigations) | 2 | 6 | 5 | 5 | 2
Haematocrit decreased (Investigations) | 2 | 2 | 4 | 0 | 0
Haemoglobin decreased (Investigations) | 2 | 2 | 3 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 2 | 3 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 1 | 3 | 3 | 1
Hypertension (Vascular disorders) | 5 | 5 | 5 | 6 | 5
Intraocular pressure increased (Investigations) | 1 | 6 | 6 | 5 | 2 — Study eye
Macular oedema (Eye disorders) | 3 | 1 | 0 | 0 | 0
Maculopathy (Eye disorders) | 2 | 2 | 1 | 4 | 3 — Study eye
Nasopharyngitis (Infections and infestations) | 4 | 4 | 3 | 1 | 3
Nausea (Gastrointestinal disorders) | 1 | 2 | 3 | 4 | 4
Ocular hyperaemia (Eye disorders) | 2 | 5 | 2 | 3 | 3 — Study eye
Oedema peripheral (General disorders) | 3 | 1 | 1 | 2 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1 | 1 | 0
Posterior capsule opacification (Eye disorders) | 3 | 1 | 1 | 1 | 0
Protein urine present (Investigations) | 2 | 1 | 1 | 4 | 3
Punctate keratitis (Eye disorders) | 1 | 1 | 0 | 3 | 0 — Study eye
Red blood cell count decreased (Investigations) | 0 | 1 | 3 | 0 | 1
Retinal aneurysm (Eye disorders) | 0 | 1 | 0 | 3 | 1
Retinal haemorrhage (Eye disorders) | 3 | 1 | 1 | 3 | 5
Retinal haemorrhage (Eye disorders) | 2 | 0 | 3 | 1 | 4 — Study eye
Retinal aneurysm (Eye disorders) | 1 | 3 | 0 | 2 | 2 — Study eye
Retinal neovascularisation (Eye disorders) | 1 | 0 | 2 | 1 | 3
Retinal exudates (Eye disorders) | 1 | 4 | 1 | 2 | 3 — Study eye
Vision blurred (Eye disorders) | 1 | 4 | 0 | 0 | 2 — Study eye
Vitreous detachment (Eye disorders) | 3 | 2 | 1 | 4 | 0
Vitreous detachment (Eye disorders) | 5 | 3 | 3 | 3 | 0 — Study eye
Vitreous floaters (Eye disorders) | 1 | 0 | 3 | 2 | 0
Vitreous floaters (Eye disorders) | 2 | 5 | 3 | 2 | 2 — Study eye
Vitreous haemorrhage (Eye disorders) | 5 | 3 | 5 | 4 | 3
Vitreous haemorrhage (Eye disorders) | 5 | 0 | 2 | 1 | 1 — Study eye

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Not less than 45 days prior to submission of a publication (S)ponsor shall be provided with a copy of the publication. The parties shall discuss any comments submitted by S regarding content, & Institution & PI shall delete any confidential information that S requests to be deleted. In addition, since the study is being conducted at multiple sites, parties agreed that publication of results shall be made only as part of a publication of the results obtained by all sites performing the study.